CLINICAL TRIAL: NCT04153019
Title: PSYCHO-EDUCATIONAL AND REHABILITATIVE INTERVENTION FOR THE ONCOLOGICAL PATIENT WITH CACHEXIA AND HIS CAREGIVER: A FEASIBILITY STUDY
Brief Title: PSYCHO-EDUCATIONAL AND REHABILITATIVE INTERVENTION FOR CANCER CACHEXIA (PRICC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AziendaUSLRE
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2023-10

CONDITIONS: Cancer Cachexia
Keywords: cancer cachexia; psychoeducational intervention; rehabilitative intervention; dyad; palliative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer cachexia (Other): Psycho-educational session: 3 weekly face-to-face consultations between a dyads (patients-caregivers) and trained nurses, helping them to cope with cancer cachexia strengthening dyadic coping resources; 2) Rehabilitation program: 3 sessions with physiotherapists including educational component for patients self-management on physical activity and goal-setting, personalized program of exercises stretching and relaxation + 3 home sessions per week, self-managed by dyads.
  Interventions: Other: Psychoeducational and rehabilitative intervention

INTERVENTIONS:
Other: Psychoeducational and rehabilitative intervention — Psycho-educational session: 3 weekly face-to-face consultations between a dyads and trained nurses, helping them to cope with cancer cachexia strengthening dyadic coping resources; 2) Rehabilitation program: 3 sessions with physiotherapists including educational component for patients self-management on physical activity and goal-setting, personalized program of exercises stretching and relaxation + 3 home sessions per week, self-managed by dyads.

SUMMARY:
Half of all cancer patients experience cachexia, with the prevalence rising above 80% in the last weeks of life. The cancer cachexia is a complex relational experience which involves the dyads patients-families. There are no studies on psychosocial interventions on dyads associated with rehabilitative interventions, to support more functional relationships to the management of cancer cachexia.

Primary objective: to evaluate the feasibility of a psycho-educational intervention combined with a physiotherapy intervention on the dyads. Secondary objective: improvement of the Quality of Life of dyads, acceptability of the intervention, adherence to each of the two components.

Methods: non-pharmacological interventional perspective, mixed-method study, addressed to a consecutive 30 cancer patients with cachexia and irreversible cachexia and their caregivers assisted by Hospital Palliative Care Unit.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Good command of the Italian language
* Written informed consent
* Histologically confirmed tumor diagnosis
* Presence of irreversible cachexia and cachexia (ESPEN3-5 guidelines, MUST calculation)
* Patients who have identified a caregiver
* Patients and family members are informed of the diagnosis and the objectives of the therapies and who have reported awareness of the disease phase (evaluated by the palliative doctor).

Exclusion Criteria:

* Patients with prognosis less than three months to enable the rehabilitative intervention
* Presence of important mental disorder or dementia
* Severe sensory deficit
* Presence of diffuse bone metastases that put the patient at risk of fracture during rehabilitation exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | After 2 months
  The proportion of number of dyads who completed the intervention / involved dyads will be evaluated. Compliance will be assessed for each individual component (psycho-social and rehabilitative intervention). The overall intervention will be evaluated feasible if there is compliance greater than or equal to 50 percent to both interventions.

SECONDARY OUTCOMES:
Functional Assessment of Anorexia-Cachexia Therapy (FAACT) | After 1 months
  Evaluation of anorexia-cachexia related distress. Each item is scored 0-4 (0=Not at all; 4= Very much). Higher scores indicating greater quality of life.
Zarit Burden Interview (ZBI) | After 1 months
  Measurement of the caregiver's perceived burden of providing family. Each item is scored 0-4 (0=Never; 4=Nearly always). Total score ranging: 0-88. Higher scores indicating greater burden.
Hand-Grip Strenght Test | After 2 months
  Measurement of isometric muscle strength of the patient's upper limbs. The best out of three attempts is accounted for.
30 seconds sit-to stand test | After 2 months
  Evaluation of functionally the strength of the lower limbs. The test counts the number of times the patient can get up from a chair without arms within a period of 30 second.
Ad-hoc semi-structured interviews aimed at the dyad | After 2 months
  Qualitative evaluation of the perception of the benefits, good adherence to the intervention or difficulties.
Ad hoc semi-structured interviews with nurses and physiotherapists | After 2 months
  Qualitative evaluation of the perception of the benefits or difficulties during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Loredana Buonaccorso, Dr., Principal Investigator — Psycho-Oncology Unit, Azienda USL - IRCSS Reggio Emilia
Locations (1):
- Loredana Buonaccorso, Reggio Emilia, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buonaccorso L, Bertocchi E, Autelitano C, Allisen Accogli M, Denti M, Fugazzaro S, Martucci G, Costi S, Tanzi S. Psychoeducational and rehabilitative intervention to manage cancer cachexia (PRICC) for patients and their caregivers: protocol for a single-arm feasibility trial. BMJ Open. 2021 Mar 1;11(3):e042883. doi: 10.1136/bmjopen-2020-042883. PMID 33649057
- [Result] Buonaccorso L, Fugazzaro S, Autelitano C, Bertocchi E, Accogli MA, Denti M, Costi S, Martucci G, Braglia L, Bassi MC, Tanzi S. Psycho-Educational and Rehabilitative Intervention to Manage Cancer Cachexia (PRICC) for Advanced Patients and Their Caregivers: Lessons Learned from a Single-Arm Feasibility Trial. Cancers (Basel). 2023 Mar 30;15(7):2063. doi: 10.3390/cancers15072063. PMID 37046724
- See also: Psychoeducational and rehabilitative intervention to manage cancer cachexia (PRICC) for patients and their caregivers: protocol for a single-arm feasibility trial — https://bmjopen.bmj.com/content/11/3/e042883

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04153019/Prot_SAP_000.pdf